CLINICAL TRIAL: NCT00422396
Title: Effects of Micronized Fenofibrate on Fasting and Postprandial Lipoproteins, Inflammatory Mediators and Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 877-017
Record Dates: First submitted 2007-01-12; First posted 2007-01-17 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Hypertriglyceridemia With the Metabolic Syndrome
Keywords: Hypertrigliceridemia; Metabolic syndrome; Obesity; Fenofibrate; Lipoproteins; Cytokines
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — Fenofibrate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Fenofibrate (drug)

SUMMARY:
This is a randomized placebo controlled clinical trial designed to investigate the effects of micronized fenofibrate on fasting and postprandial lipoproteins, oxidized fatty acids and lipoproteins, inflammatory mediators and thrombotic factors among hypertriglyceridemic individuals with two or more other characteristics of the metabolic syndrome.

DETAILED DESCRIPTION:
The aim of this study was to determine the effects of micronized fenofibrate (160 mg/daily) on:

1. Fasting and postprandial lipids and lipoproteins after a standarized test meal.
2. Fasting and postprandial oxidized fatty acids and oxidized low density lipoprotein after a standarized test meal.
3. Fasting and postprandial inflammatory mediators after a standarized test meal.
4. Fasting and postprandial lipopolysaccharide-stimulated cytokine production after a standarized test meal.
5. Fasting and postprandial markers of hemostasis, fibrinolysis and blood viscosity after a standarized test meal.

ELIGIBILITY:
Inclusion Criteria:

1. males and postmenopausal females 18 years of age with fasting triglycerides greater than or equal to 1.7 mmol/L and <6.9 mmol/L
2. two or more of the following Adult Treatment Panel III (1) criteria of the metabolic syndrome: abdominal obesity (waist circumference >89 cm in females and >102 cm in males); low high-density lipoprotein cholesterol (HDL-C) (<1.3 mmol/L in women and <1.0 mmol/L in men); hypertension (systolic blood pressure >130 or diastolic blood pressure >85 mm Hg) or current drug therapy for hypertension; and impaired fasting glucose (between 6.1 mmol/L and 7.0 mmol/L).

Exclusion Criteria:

1. included types 1 or 2 diabetes
2. Body mass index >40 kg/m2
3. Use of lipid-lowering therapies
4. Oral hypoglycemic therapies
5. Insulin
6. Aspirin >81 mg daily
7. Regular use of non-steroidal anti-inflammatory agents or cyclooxygenase-2 inhibitors, corticosteroids (oral and inhaled), anti-oxidants (including multivitamins), herbal or fiber supplements recent changes in type or formulation of hormone replacement therapy (in the last 6 months)
8. Alcohol intake >3 drinks per day
9. Untreated hypothyroidism or recent change (within 2 months) of thyroid replacement therapy
10. Cigarette smoking (current or within the last 6 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2001-01 (Actual); Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
1. lipids and lipoproteins

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Rosenson, MD, Principal Investigator — University of Michigan
Locations (1):
- Northwestern University preventive Cardiology Center, Chicago, Illinois, United States